CLINICAL TRIAL: NCT02499016
Title: Suprapubic Single-incision Laparoscopic Appendectomy Versus Conventional Multiport Appendectomy: a Randomized Controlled Trial
Brief Title: Suprapubic Single-incision Laparoscopic Appendectomy Versus Conventional Appendectomy: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFGS-SSILA-01
Record Dates: First submitted 2015-06-10; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-03

CONDITIONS: Complications
Keywords: Appendicitis; Appendectomy; Single-incision
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- suprapubic single-incision laparoscopic appendectomy (Experimental): single incision laparoscopic surgery will be performed for patients in this group.
  Interventions: Procedure: suprapubic single-incision laparoscopic appendectomy
- conventional multiport appendectomy (Active Comparator): Conventional laparoscopic surgery will be performed for patients in this group.
  Interventions: Procedure: suprapubic single-incision laparoscopic appendectomy

INTERVENTIONS:
Procedure: suprapubic single-incision laparoscopic appendectomy — the approach of appendectomy
  Other Names: SSILA

SUMMARY:
Conventional laparoscopic appendectomy(CLA) is the current standard treatment. To obtain additional benefits such as a better cosmetic outcome, the investigators developed a surgical option termed suprapubic single-incision laparoscopic appendectomy (SSILA), which creates a non-visible scar, that was preliminarily shown to be feasible and safe in our previous retrospective studies To further evaluate the feasibility, safety and cosmetic results of this innovative approach, the investigators compared the outcomes of SSILA and CLA by performing a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* acute appendicitis or interval appendicitis
* informed consent

Exclusion Criteria:

* diagnosis of appendicitis was not clinically established (symptoms attributable to urinary or gynecological problems)
* history of cirrhosis and coagulation disorders
* suspected or proven malignancy
* contraindication to general anesthesia (severe cardiac and/or pulmonary disease)
* inability to give informed consent(severe mental disease)
* pregnancy
* BMI>30kg/m2
* generalized peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
incidence of complications | 30 days
  The early morbidity rate is defined as the event observed during operation and within 30 days after surgery

SECONDARY OUTCOMES:
mortality rate | 30 days
cosmetic results | 30 days
  Cosmetic assessment is perform using body image scale and cosmetic scale.
operative time | intraoperative
time to recover | 14 days
Pain score | 14 days
  Postoperative pain is recorded using the visual analog scale (VAS) pain score tool on postoperative day 1, 2, 3 and the day of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, M.D.,Ph. D., Principal Investigator — Nanfang Hospital, Southern Medical University, China
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Yu J, Wang YN, Hu YF, Cheng X, Zhen L, Li GX. Single-incision laparoscopic appendectomy performed above the pubic symphysis - a new scarless approach. Minim Invasive Ther Allied Technol. 2011 Jan;20(1):18-21. doi: 10.3109/13645706.2010.518672. PMID 21222504
- [Result] Wang Y, Xiong W, Lan X, Zhang J, Chen T, Liu H, Li G. Suprapubic single incision laparoscopic appendectomy. J Surg Res. 2015 Feb;193(2):577-82. doi: 10.1016/j.jss.2014.07.064. Epub 2014 Aug 4. PMID 25179807